CLINICAL TRIAL: NCT02312921
Title: Reducing Oral Health Disparity Through Outreach, Evidenced-Based Care, Global Budgeting and the Alternative Quality Contract
Brief Title: Population-centered Risk- and Evidence-based Dental Inter-professional Care Team
Acronym: PREDICT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Advantage Dental Services, LLC (Industry)
Collaborators: Robert Wood Johnson Foundation (Other); University of Chicago (Other); University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: RWJF
Record Dates: First submitted 2014-12-06; First posted 2014-12-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Dental Caries
Keywords: managed healthcare; child; dental care
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PREDICT: Delivery system changes where a team of dental providers (dentists, dental hygienists, case managers, community outreach workers and others) within Advantage Dental Services, LLC provide evidence-based screening, risk assessment and primary and secondary preventive care in non-conventional community settings (WIC, Head Start and similar settings) and seamless, timely and appropriate evidence-based care in dental clinics.
  Payment plan model based on global budgeting and Alternative Quality Contract (pay-for-performance) for dental providers within Advantage Dental Services, LLC (Advantage) with the goal of incentivizing implementation of delivery system changes aimed at reducing disparities in dental care utilization and oral health for low-income mothers and children..
  Interventions: Other: PREDICT
- Control: Usual care

INTERVENTIONS:
Other: PREDICT — Allied dental personnel provide screening and preventive services in community settings and case managers serve as patient navigators to arrange referrals of children who need dentist services. The intervention is paired with a compensation system for high performance (pay-for-performance) with efficient performance monitoring. PREDICT focuses on: 1) identifying eligible children and gaining caregiver consent for services in community settings (e.g., schools); 2) providing risk-based preventive and caries stabilization services efficiently at these settings; 3) providing curative care in dental clinics; and 4) incentivizing local delivery teams to meet performance benchmarks.
  Groups: PREDICT

SUMMARY:
The main goal of the payment and delivery system reform is to reduce disparities in oral health and dental care access of low-income mothers and children living in rural Oregon counties. The target population is children, pregnant women and new mothers enrolled in Oregon Health Plan (OHP) in rural Oregon.

DETAILED DESCRIPTION:
To implement a payment plan model based on global budgeting and Alternative Quality Contract (pay-for-performance) for dental providers within Advantage Dental Services, LLC with the goal of incentivizing implementation of delivery system changes aimed at reducing disparities in access and oral health for low-income mothers and children living in rural Oregon counties.

To implement delivery system changes where a team of dental providers (dentists, dental hygienists, case managers, community outreach workers and others) within Advantage Dental Services, LLC provide evidence-based screening, risk assessment and primary preventive care in non-conventional community settings (WIC, Head Start and similar settings) and seamless, timely and appropriate evidence-based care in Advantage dental clinics.

To evaluate and document the payment and delivery system changes to assess whether the changes result in (1) reductions in disparities in access for low-income mothers and children; (2) efficiency in allocation of limited resources with the application of evidence-based screening; (3) seamless and appropriate care for mothers and their child at high risk of dental caries

ELIGIBILITY:
Inclusion Criteria:

* Children less than 21 years old and women who are pregnant or up to 2 months-post-partum.
* Enrollment in Medicaid and assigned by Oregon Health Authority to receive dental care from Advantage Dental Plan.
* Home address is located in the selected counties.

Exclusion Criteria:

* None

Max Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 80,000 children on Medicaid nested in 14 rural Oregon Counties.
Sampling Method: Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Untreated dental caries | 2 years
  Percentage of participants with untreated dental caries

SECONDARY OUTCOMES:
Consumer Satisfaction | 2 years
  Scores on the Dental Satisfaction Questionnaire
Dental care utilization | 2 years
  Percentage of participants 0-21 years of age and pregnant women who received a dental service

CONTACTS AND LOCATIONS:
Overall Officials: Peter Milgrom, DDS, Study Director — Advantage Dental Services, LLC

REFERENCES:
- [Derived] Cunha-Cruz J, Milgrom P, Shirtcliff RM, Bailit HL, Huebner CE, Conrad D, Ludwig S, Mitchell M, Dysert J, Allen G, Scott J, Mancl L. Population-centered Risk- and Evidence-based Dental Interprofessional Care Team (PREDICT): study protocol for a randomized controlled trial. Trials. 2015 Jun 20;16:278. doi: 10.1186/s13063-015-0786-y. PMID 26091669